CLINICAL TRIAL: NCT02341885
Title: PrEvalence of Acute and Chronic Kidney Disease Treated by Renal Replacement Therapy in the ICU Environment
Brief Title: PrEvalence of Acute and Chronic Kidney Disease Treated by Renal Replacement Therapy
Acronym: PEACE
Status: Completed | Type: Observational
Sponsor: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: PEACE
Record Dates: First submitted 2015-01-12; First posted 2015-01-19 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Renal Replacement Therapy; Acute Kidney Injury; Chronic End Stage Kidney Disease
Keywords: Kidney; Renal replacement; Acute kidney injury; chronic kidney disease; Epidemiology; Prevalence
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- One Group: This is an observational study, aimed at collecting an adequate dataset on a large cohort of patients admitted to a large number of ICUs.

SUMMARY:
A prospective international, multi-centre, prevalence study on the epidemiology of the use of renal replacement therapy for ICU patients who have acute kidney injury and chronic end stage kidney disease.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common finding in intensive care unit (ICU) patients. Approximately 30 to 65% of patients experience an episode of AKI, and 5% of ICU patients are treated with renal replacement therapy. AKI is associated withimportant short term and long-term morbidity as well as mortality, and therefore also with costs. Finally, there is a close link between chronic kidney disease (CKD) and AKI. CKD patients are at greater risk for developing AKI, and survivors of AKI treated with renal replacement therapy (AKI-RRT), may develop chronic kidney disease (CKD) and end stage kidney disease (ESKD).

Different aspects of RRT modality may impact on outcomes, and data that have emerged over the last decade have improved evidence and also rejected commonly accepted dogma. Initial data suggested a better outcome when a higher dose of treatment was applied [5,6]. However, one small and two large prospective randomised controlled trials failed to reproduce these earlier findings. Observational data seems to suggest that continuous RRT (CRRT) modalities are associated with better outcomes. However, relative small, randomized studies and meta-analyses do not demonstrate such a benefit. Observational data suggests that CRRT is associated with improved renal recovery, and also examining the data from the 2 large randomized studies on intensity of RRT suggest that CRRT confers a benefit. Also, despite RRT being available for over 50 years there are no clear consensus guidelines for the initiation of RRT. A recent survey found that up to 89 different combinations of indications are used. Recently, the Acute Kidney Injury Network and the Kidney Disease: Improving Global Outcomes (KDIGO) group, formulated recommendations for this. Recent observational studies indicated that commonly accepted cut offs such as serum urea concentration are probably not that important. Furthermore, timing of initiation may have an effect on outcome. Some studies suggest that early initiation is associated with better outcome, on the other hand others could not demonstrate a benefit and have even demonstrated inferior outcomes.

The most recent survey in Europe showed that CRRT is the preferred modality among intensivists, and that despite the recently published evidence treatment doses are similar to those of a decade ago.

Data on the use of renal replacement therapy (RRT) for AKI and for CKD in ICU patients are either on specific patient groups, such as cardiac surgery patients, based on surveys, or dates back for at least a decade. Furthermore, these studies suffered from exclusion bias, as patients who fulfilled criteria for initiation of RTT, but who were denied RRT, were not considered. That this may be an important consideration is illustrated by findings from a recent small single centre study that demonstrated similar mortality rate between RIFLE-F patients who were and who were not treated with RRT. Therefore, the Acute Kidney Injury Network (AKIN) recommended measuring the epidemiology of AKI.

The investigators anticipate that the evidence that has been generated on different topics of RRT for ICU patients may have influenced current practice. Also, the investigators anticipate regional differences in RRT practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients present in the ICU at time of the study data (date starting at 0:00 h, and ending at 23:59 h) (index ICU stay)
* ≥18 years of age
* When required by local EC regulations and EC approval, informed consent (written or oral) by the patient or relative.

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care Unit patients diagnosed with acute kidney injury and chronic end stage kidney disease.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of severe AKI | with a maximum follow up till day 28 following the index study day
  Assessment of the prevalence of severe AKI (defined as KDIGO class 3) and CKD (defined by treatment with renal replacement therapy (RRT)), in ICU patients, present at time of the study inclusion day

SECONDARY OUTCOMES:
Modalities of RRT | with a maximum follow up till day 28 following the index study day
  Assessment of modalities of RRT used for treatment of AKI
Indications for initiation of RRT | with a maximum follow up till day 28 following the index study day
  Assessment of indications for initiation of RRT currently described in literature
Severity of illness | with a maximum follow up till day 28 following the index study day
  Assessment of severity of illness at time of data recording
Renal outcome | with a maximum follow up till day 28 following the index study day
  Assessment of renal outcome

CONTACTS AND LOCATIONS:
Overall Officials: Eric HOSTE, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- All Centres From All Over the World Willing to Contribute Are Welcome, Brussels, Belgium

REFERENCES:
- [Background] Metnitz PG, Krenn CG, Steltzer H, Lang T, Ploder J, Lenz K, Le Gall JR, Druml W. Effect of acute renal failure requiring renal replacement therapy on outcome in critically ill patients. Crit Care Med. 2002 Sep;30(9):2051-8. doi: 10.1097/00003246-200209000-00016. PMID 12352040
- [Background] Uchino S, Kellum JA, Bellomo R, Doig GS, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Ronco C; Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) Investigators. Acute renal failure in critically ill patients: a multinational, multicenter study. JAMA. 2005 Aug 17;294(7):813-8. doi: 10.1001/jama.294.7.813. PMID 16106006
- [Background] Hoste EA, Schurgers M. Epidemiology of acute kidney injury: how big is the problem? Crit Care Med. 2008 Apr;36(4 Suppl):S146-51. doi: 10.1097/CCM.0b013e318168c590. PMID 18382186
- [Background] Hoste EAJ, J.A. K, group TAKI-EPIs: The epidemiology of acute kidney injury - Preliminary results of the multicenter international AKI-EPI study. Intensive Care Med 2011, 37: S207
- [Background] Ronco C, Bellomo R, Homel P, Brendolan A, Dan M, Piccinni P, La Greca G. Effects of different doses in continuous veno-venous haemofiltration on outcomes of acute renal failure: a prospective randomised trial. Lancet. 2000 Jul 1;356(9223):26-30. doi: 10.1016/S0140-6736(00)02430-2. PMID 10892761
- [Background] Schiffl H, Lang SM, Fischer R. Daily hemodialysis and the outcome of acute renal failure. N Engl J Med. 2002 Jan 31;346(5):305-10. doi: 10.1056/NEJMoa010877. PMID 11821506
- [Background] Bouman CS, Oudemans-Van Straaten HM, Tijssen JG, Zandstra DF, Kesecioglu J. Effects of early high-volume continuous venovenous hemofiltration on survival and recovery of renal function in intensive care patients with acute renal failure: a prospective, randomized trial. Crit Care Med. 2002 Oct;30(10):2205-11. doi: 10.1097/00003246-200210000-00005. PMID 12394945
- [Background] VA/NIH Acute Renal Failure Trial Network; Palevsky PM, Zhang JH, O'Connor TZ, Chertow GM, Crowley ST, Choudhury D, Finkel K, Kellum JA, Paganini E, Schein RM, Smith MW, Swanson KM, Thompson BT, Vijayan A, Watnick S, Star RA, Peduzzi P. Intensity of renal support in critically ill patients with acute kidney injury. N Engl J Med. 2008 Jul 3;359(1):7-20. doi: 10.1056/NEJMoa0802639. Epub 2008 May 20. PMID 18492867
- [Background] RENAL Replacement Therapy Study Investigators; Bellomo R, Cass A, Cole L, Finfer S, Gallagher M, Lo S, McArthur C, McGuinness S, Myburgh J, Norton R, Scheinkestel C, Su S. Intensity of continuous renal-replacement therapy in critically ill patients. N Engl J Med. 2009 Oct 22;361(17):1627-38. doi: 10.1056/NEJMoa0902413. PMID 19846848
- [Background] Forni LG, Hilton PJ. Continuous hemofiltration in the treatment of acute renal failure. N Engl J Med. 1997 May 1;336(18):1303-9. doi: 10.1056/NEJM199705013361807. No abstract available. PMID 9113935
- [Background] Mehta RL, McDonald B, Gabbai FB, Pahl M, Pascual MT, Farkas A, Kaplan RM; Collaborative Group for Treatment of ARF in the ICU. A randomized clinical trial of continuous versus intermittent dialysis for acute renal failure. Kidney Int. 2001 Sep;60(3):1154-63. doi: 10.1046/j.1523-1755.2001.0600031154.x. PMID 11532112
- [Background] Vinsonneau C, Camus C, Combes A, Costa de Beauregard MA, Klouche K, Boulain T, Pallot JL, Chiche JD, Taupin P, Landais P, Dhainaut JF; Hemodiafe Study Group. Continuous venovenous haemodiafiltration versus intermittent haemodialysis for acute renal failure in patients with multiple-organ dysfunction syndrome: a multicentre randomised trial. Lancet. 2006 Jul 29;368(9533):379-85. doi: 10.1016/S0140-6736(06)69111-3. PMID 16876666
- [Background] Lins RL, Elseviers MM, Van der Niepen P, Hoste E, Malbrain ML, Damas P, Devriendt J; SHARF investigators. Intermittent versus continuous renal replacement therapy for acute kidney injury patients admitted to the intensive care unit: results of a randomized clinical trial. Nephrol Dial Transplant. 2009 Feb;24(2):512-8. doi: 10.1093/ndt/gfn560. Epub 2008 Oct 14. PMID 18854418
- [Background] Uehlinger DE, Jakob SM, Ferrari P, Eichelberger M, Huynh-Do U, Marti HP, Mohaupt MG, Vogt B, Rothen HU, Regli B, Takala J, Frey FJ. Comparison of continuous and intermittent renal replacement therapy for acute renal failure. Nephrol Dial Transplant. 2005 Aug;20(8):1630-7. doi: 10.1093/ndt/gfh880. Epub 2005 May 10. PMID 15886217
- [Background] Bagshaw SM, Berthiaume LR, Delaney A, Bellomo R. Continuous versus intermittent renal replacement therapy for critically ill patients with acute kidney injury: a meta-analysis. Crit Care Med. 2008 Feb;36(2):610-7. doi: 10.1097/01.CCM.0B013E3181611F552. PMID 18216610
- [Background] Pannu N, Klarenbach S, Wiebe N, Manns B, Tonelli M; Alberta Kidney Disease Network. Renal replacement therapy in patients with acute renal failure: a systematic review. JAMA. 2008 Feb 20;299(7):793-805. doi: 10.1001/jama.299.7.793. PMID 18285591
- [Background] Bell M, Granath F, Schon S, Lofberg E; SWING; Ekbom A, Martling CR. End-stage renal disease patients on renal replacement therapy in the intensive care unit: short- and long-term outcome. Crit Care Med. 2008 Oct;36(10):2773-8. doi: 10.1097/CCM.0b013e318187815a. PMID 18766088
- [Background] Bell M; SWING; Granath F, Schon S, Ekbom A, Martling CR. Continuous renal replacement therapy is associated with less chronic renal failure than intermittent haemodialysis after acute renal failure. Intensive Care Med. 2007 May;33(5):773-780. doi: 10.1007/s00134-007-0590-6. Epub 2007 Mar 16. PMID 17364165
- [Background] Uchino S, Bellomo R, Kellum JA, Morimatsu H, Morgera S, Schetz MR, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Oudemans-Van Straaten HM, Ronco C; Beginning and Ending Supportive Therapy for the Kidney (B.E.S.T. Kidney) Investigators Writing Committee. Patient and kidney survival by dialysis modality in critically ill patients with acute kidney injury. Int J Artif Organs. 2007 Apr;30(4):281-92. doi: 10.1177/039139880703000402. PMID 17520564
- [Background] Ricci Z, Ronco C, D'Amico G, De Felice R, Rossi S, Bolgan I, Bonello M, Zamperetti N, Petras D, Salvatori G, Dan M, Piccinni P. Practice patterns in the management of acute renal failure in the critically ill patient: an international survey. Nephrol Dial Transplant. 2006 Mar;21(3):690-6. doi: 10.1093/ndt/gfi296. Epub 2005 Dec 2. PMID 16326743
- [Background] Gibney N, Hoste E, Burdmann EA, Bunchman T, Kher V, Viswanathan R, Mehta RL, Ronco C. Timing of initiation and discontinuation of renal replacement therapy in AKI: unanswered key questions. Clin J Am Soc Nephrol. 2008 May;3(3):876-80. doi: 10.2215/CJN.04871107. Epub 2008 Mar 5. PMID 18322044
- [Background] Ostermann M, Chang RW. Correlation between parameters at initiation of renal replacement therapy and outcome in patients with acute kidney injury. Crit Care. 2009;13(6):R175. doi: 10.1186/cc8154. Epub 2009 Nov 4. PMID 19889205
- [Background] De Corte W, Vanholder R, Dhondt AW, De Waele JJ, Decruyenaere J, Danneels C, Claus S, Hoste EA. Serum urea concentration is probably not related to outcome in ICU patients with AKI and renal replacement therapy. Nephrol Dial Transplant. 2011 Oct;26(10):3211-8. doi: 10.1093/ndt/gfq840. Epub 2011 Mar 18. PMID 21421593
- [Background] Bouman CS, Forni LG. Initiation of renal replacement therapy: is timing everything? Crit Care. 2010;14(1):107. doi: 10.1186/cc8188. Epub 2010 Feb 10. PMID 20236445
- [Background] Bagshaw SM, Uchino S, Bellomo R, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Oudemans-van Straaten HM, Ronco C, Kellum JA; Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) Investigators. Timing of renal replacement therapy and clinical outcomes in critically ill patients with severe acute kidney injury. J Crit Care. 2009 Mar;24(1):129-40. doi: 10.1016/j.jcrc.2007.12.017. Epub 2008 Apr 18. PMID 19272549
- [Background] Seabra VF, Balk EM, Liangos O, Sosa MA, Cendoroglo M, Jaber BL. Timing of renal replacement therapy initiation in acute renal failure: a meta-analysis. Am J Kidney Dis. 2008 Aug;52(2):272-84. doi: 10.1053/j.ajkd.2008.02.371. Epub 2008 Jun 18. PMID 18562058
- [Background] Kumpers P, Hafer C, Lukasz A, Lichtinghagen R, Brand K, Fliser D, Faulhaber-Walter R, Kielstein JT. Serum neutrophil gelatinase-associated lipocalin at inception of renal replacement therapy predicts survival in critically ill patients with acute kidney injury. Crit Care. 2010;14(1):R9. doi: 10.1186/cc8861. Epub 2010 Feb 1. PMID 20122150
- [Background] Vinsonneau C, Monchi M. Too early initiation of renal replacement therapy may be harmful. Crit Care. 2011;15(1):112. doi: 10.1186/cc9405. Epub 2011 Jan 26. PMID 21345253
- [Background] Legrand M, Darmon M, Joannidis M, Payen D. Management of renal replacement therapy in ICU patients: an international survey. Intensive Care Med. 2013 Jan;39(1):101-8. doi: 10.1007/s00134-012-2706-x. Epub 2012 Sep 22. PMID 23001448
- [Background] Bell M, Liljestam E, Granath F, Fryckstedt J, Ekbom A, Martling CR. Optimal follow-up time after continuous renal replacement therapy in actual renal failure patients stratified with the RIFLE criteria. Nephrol Dial Transplant. 2005 Feb;20(2):354-60. doi: 10.1093/ndt/gfh581. Epub 2004 Dec 14. PMID 15598666
- [Background] Ronco C, Ricci Z, Bellomo R. Current worldwide practice of dialysis dose prescription in acute renal failure. Curr Opin Crit Care. 2006 Dec;12(6):551-6. doi: 10.1097/01.ccx.0000247447.17124.05. PMID 17077685
- [Background] Uchino S, Bellomo R, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Oudemans-van Straaten H, Ronco C, Kellum JA. Continuous renal replacement therapy: a worldwide practice survey. The beginning and ending supportive therapy for the kidney (B.E.S.T. kidney) investigators. Intensive Care Med. 2007 Sep;33(9):1563-70. doi: 10.1007/s00134-007-0754-4. Epub 2007 Jun 27. PMID 17594074
- [Background] Mehta RL, Pascual MT, Soroko S, Savage BR, Himmelfarb J, Ikizler TA, Paganini EP, Chertow GM; Program to Improve Care in Acute Renal Disease. Spectrum of acute renal failure in the intensive care unit: the PICARD experience. Kidney Int. 2004 Oct;66(4):1613-21. doi: 10.1111/j.1523-1755.2004.00927.x. PMID 15458458
- [Background] Kellum JA, Mehta RL, Levin A, Molitoris BA, Warnock DG, Shah SV, Joannidis M, Ronco C; Acute Kidney Injury Network (AKIN). Development of a clinical research agenda for acute kidney injury using an international, interdisciplinary, three-step modified Delphi process. Clin J Am Soc Nephrol. 2008 May;3(3):887-94. doi: 10.2215/CJN.04891107. Epub 2008 Jan 23. PMID 18216348
- [Background] Cerda J, Lameire N, Eggers P, Pannu N, Uchino S, Wang H, Bagga A, Levin A. Epidemiology of acute kidney injury. Clin J Am Soc Nephrol. 2008 May;3(3):881-6. doi: 10.2215/CJN.04961107. Epub 2008 Jan 23. PMID 18216347
- [Background] Vaara ST, Korhonen AM, Kaukonen KM, Nisula S, Inkinen O, Hoppu S, Laurila JJ, Mildh L, Reinikainen M, Lund V, Parviainen I, Pettila V; FINNAKI Study Group. Fluid overload is associated with an increased risk for 90-day mortality in critically ill patients with renal replacement therapy: data from the prospective FINNAKI study. Crit Care. 2012 Oct 17;16(5):R197. doi: 10.1186/cc11682. PMID 23075459
- [Background] Davenport A. Clinical guidelines for the protection of kidney function and prevention of acute kidney injury in the intensive care unit: common sense rather than magic bullets? Intensive Care Med. 2010 Mar;36(3):379-80. doi: 10.1007/s00134-009-1683-1. No abstract available. PMID 19921151